CLINICAL TRIAL: NCT01732731
Title: Effects of Intensive Locomotor Treadmill Training on Gross Motor Function in Young Children With Neuromotor Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-97; 527109 (Other Grant/Funding Number: Am PhysTherapy Assoc. Pediatric Research Grant 527109)
Record Dates: First submitted 2012-09-24; First posted 2012-11-26 (Estimated); Last update posted 2012-11-26 (Estimated); Status verified 2012-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; treadmill training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treadmill training (Experimental): children will receive home-based treadmill training with supervision from a physical therapist
  Interventions: Other: treadmill training
- no treadmill training (No Intervention): children will not receive treadmill training

INTERVENTIONS:
Other: treadmill training — Home-based treadmill training will be administered to the children in the experimental group
  Arms: treadmill training

SUMMARY:
The purpose of this project is to examine if early exposure to intensive, short-term locomotor treadmill training (LT) in young children with neuromotor impairment will help develop walking skills earlier, decrease the amount of outside assistance needed (such as a walker or crutches) as compared to children with neuromotor impairment who receive traditional physical therapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of CP with GMFCS levels I and II
* ages 9 to 36 months
* the ability to sit for at least 30 seconds unsupported in ring-sitting or W-sitting
* the ability to take ten consecutive steps when held on hands

Exclusion Criteria:

* a diagnosis of a genetic syndrome
* independent ambulation without an assistive device
* previous or current use of treadmill intervention during physical therapy
* a medical contraindication for standing or walking defined by the physician 5) uncontrolled seizures
* a history of orthopedic surgery
* use of medication to control spasticity in the past 6 months

Ages: 9 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure Dimension D and E | up to 4-months post-intervention

SECONDARY OUTCOMES:
Peabody Developmental Motor Scales-2 | pre-intervention, 6-week post-intervention, 1-month post-intervention, 4-month post-intervention
timed 10 meter walk test | pre-intervention, 6-week post-intervention, 1-month post-intervention, 4-month post-intervention
Pediatric Evaluation of Disability Inventory | pre-intervention, 6-week post-intervention, 1-month post-intervention, 4-month post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Mattern-Baxter, Principal Investigator — University of the Pacific